CLINICAL TRIAL: NCT02264002
Title: Pharmacodynamic Effects, Safety and Tolerability of 0.25 mg, 0.5 mg, 1 mg and 2 mg Cilobradine, Compared to 190 mg Metoprolol Succinate and Placebo, Administered p.o. Once Daily Over 14 Days to Healthy Volunteers in a Randomised, Placebo-controlled, Partly Double Blind Study, With a 4 mg/14 mg and 10 mg/20 mg Cilobradine Single Dose Versus Placebo Substudy (Double Blind, Three-fold Cross-over)
Brief Title: Pharmacodynamic Effects, Safety and Tolerability of Cilobradine, Compared to Metoprolol Succinate and Placebo in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 503.203
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — cilobradine; Metoprolol

ARMS (7):
- Cilobradine low dose 1 (Experimental)
  Interventions: Drug: Cilobradine low dose 1
- Cilobradine low dose 2 (Experimental)
  Interventions: Drug: Cilobradine low dose 2
- Cilobradine medium dose (Experimental)
  Interventions: Drug: Cilobradine medium dose
- Cilobradine high dose 1 (Experimental)
  Interventions: Drug: Cilobradine high dose 1
- Cilobradine high dose 2 (Experimental)
  Interventions: Drug: Cilobradine high dose 2
- Metoprolol succinate (Active Comparator): 1 tablet on day 1, day 2 followed by two tablets from day 3 to day 14
  Interventions: Drug: Metoprolol succinate tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilobradine low dose 1
  Arms: Cilobradine low dose 1
Drug: Cilobradine low dose 2
  Arms: Cilobradine low dose 2
Drug: Cilobradine medium dose
  Arms: Cilobradine medium dose
Drug: Cilobradine high dose 1
  Arms: Cilobradine high dose 1
Drug: Cilobradine high dose 2
  Arms: Cilobradine high dose 2
Drug: Metoprolol succinate tablets
  Arms: Metoprolol succinate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Pharmacodynamic effects on heart rate (HR) at rest and during exercise and on flicker fusion frequency (FFF), FFF method evaluation

Safety, tolerability and pharmacokinetics of cilobradine

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males and females. Volunteers will

  * be 21 to 55 years of age
  * have a Body Mass Index (BMI) of 19.9 to 29.9 kg/m2 and
  * have a resting heart rate (HR) (after 10 min. in the supine position) of more than 55 beats per minute (bpm)
* Only post-menopausal females, or those who had had a hysterectomy, could participate. All females had to have a negative pregnancy test
* In accordance with good clinical practice (GCP) and the local legislation all volunteers had to give their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including BP, HR and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the Investigator
* Intake of drugs with a long half-life (> 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial within two weeks prior to administration or during the trial
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 ml within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Not necessarily clinically relevant abnormalities, but specific Exclusion criteria for the drugs under study or for the study:

* Consumption of more than 2 cups of coffee or black tea, or cola drinks, per day during the last 6 weeks. However, subjects may participate if abstinence from the before mentioned beverages is well tolerated during an interval of at least 2 weeks between screening and first treatment
* ECG: PQ interval > 210 ms
* HR at rest < 55 bpm
* Systolic BP < 115 mmHg
* Colour vision test abnormal. However, subjects may participate if they are able to perform the flicker fusion test without difficulty
* Psoriasis (own medical history or relative)
* Relevant ophthalmological disease
* History of asthma or obstructive pulmonary disease
* History (including childhood) of traumatic injury to the head or brain
* History (including childhood) of reduced seizure threshold
* The following subjects will not be allowed to participate in the study

  * Any subject involved in professional transportation of human subjects
  * Any subject involved in operating dangerous machinery

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2003-02; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate at rest | Pre-dose, up to day 20 after first drug administration
Changes in heart rate during exercise | Pre-dose, up to day 20 after first drug administration
Changes in flicker fusion frequency test (FFF) | Pre-dose, up to day 20 after first drug administration

SECONDARY OUTCOMES:
Number of patients with clinically relevant changes in laboratory tests | Pre-dose, up to 12 days after last drug administration
Number of patients with clinically relevant changes in vital signs (blood pressure, heart rate) | Pre-dose, up to 12 days after last drug administration
Number of patients with clinically relevant changes in 12-lead ECG | Pre-dose, up to 12 days after last drug administration
Number of patients with adverse events | Up to 12 days after last drug administration
Assessment of global tolerability by the investigator | Up to 12 days after last drug administration
Changes in peripheral FFF | Pre-dose, up to day 20 after first drug administration
Area under the concentration-time curve of the analytes in plasma (AUC) | Up to day 20 after start of first drug administration
Maximum measured concentration of the analytes in plasma (Cmax) | Up to day 20 after start of first drug administration
Time from dosing to the maximum concentration of the analytes in plasma (tmax) | Up to day 20 after start of first drug administration
Terminal half-life of the analytes in plasma (t½) | Up to day 20 after start of first drug administration
Mean residence time of the analytes in the body after oral administration (MRTpo) | Up to day 20 after start of first drug administration
Total clearance of the analytes in plasma following extravascular administration (CL/F) | Up to day 20 after start of first drug administration
Apparent volume of distribution of the analytes during the terminal phase λz following extravascular administration (Vz/F) | Up to day 20 after start of first drug administration